CLINICAL TRIAL: NCT02027740
Title: Effect of Almond Supplementation on Glycemic and Cardiovascular Risk Factors in Asian Indians in North India With Type 2 Diabetes Mellitus: A 24-week Prospective Cohort Study
Brief Title: Almond Intervention in Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diabetes Foundation, India (Other)
Responsible Party: Principal Investigator, Dr Anoop Misra, Director, Diabetes Foundation, India
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: almond.2013
Record Dates: First submitted 2014-01-03; First posted 2014-01-06 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- almond (Experimental): almonds are substituted for visible fat and carbohydrates
  Interventions: Dietary Supplement: almond

INTERVENTIONS:
Dietary Supplement: almond

SUMMARY:
This prospective cohort study of an almond-enriched diet (within the overall context of Asian Indian dietary guidelines) was conducted to test the hypothesis that in patients with T2DM almond-enriched balanced diet improves glycemic measures and CVD risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the age range of 25-65 years
* on stable doses of metformin from past 3 months
* having HbA1C less than 9%
* LDL-c ≥100 mg/dl were recruited

Exclusion Criteria:

* Patients on insulin therapy, plioglitazone, insulin secretagogues, beta blockers or steroids or suffering from diabetes for more than 10 years
* having high uric acid levels (≥ 8 mg/dl),
* with accelerated hypertension (stage 2 hypertension according to JNC guidelines) , hypothyroidism, suffering from acute infection or any debilitating disease or with renal failure,
* appreciable weight loss (more than 10%) during past 6 months
* Patients with known food allergy, lipid altering medication or extraneous factors that can affect glycemic or lipid parameters

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-01; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change in LDL-c | baseline, after six months

SECONDARY OUTCOMES:
HbA1C | baseline, after six months of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Fortis Flt Lt Hospital, Delhi, India